CLINICAL TRIAL: NCT03982290
Title: Psychophysiological Effects of Lactobacillus Plantarum PS128 in Preschool Children With Autism Spectrum Disorder: a Randomized, Placebo-controlled Trial
Brief Title: Psychophysiological Effects of Lactobacillus Plantarum PS128 in Preschool Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Ju Chen, Senior Attending Physician, Mackay Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17MMHIS193e
Record Dates: First submitted 2019-05-31; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Autism
Keywords: autism; preschool children
MeSH Terms: conditions — Autistic Disorder | interventions — Probiotics; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, researchers, outcome assessors, subjects and caregivers will be blinded to the randomization. A research assistant who is not involved in this trial will do the randomization by using randomly permuted blocks within the strata of two assignments, the placebo group and PS128 group with the ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus plantarum PS128 (PS128) (Active Comparator): Subjects will receive oral Lactobacillus plantarum PS128 capsules, 2 capsules per day, for 16 weeks.
  Interventions: Other: Probiotic, Lactobacillus plantarum PS128
- Placebo (Placebo Comparator): Subjects will receive oral placebo capsules, 2 capsules per day, for the first 8 weeks. The following 8 weeks, subjects will receive oral Lactobacillus plantarum PS128 capsules, 2 capsules per day, for 8 weeks.
  Interventions: Other: Placebo, microcrystalline cellulose
- Normal Control (No Intervention): Normal control group are enrolled by invitation from the age and gender matched healthy children.

INTERVENTIONS:
Other: Probiotic, Lactobacillus plantarum PS128 — PS128 capsules, 2 capsules per day
  Other Names: PS128
  Arms: Lactobacillus plantarum PS128 (PS128)
Other: Placebo, microcrystalline cellulose — Placebo capsules, 2 capsules per day
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Autism Spectrum Disorders (ASD) comprises a complex group of disorders of neuronal development characterized by social and communication impairment along with presence of repetitive and restrictive behaviors. Emerging evidences support the gut-brain axis and further microbiota-gut-brain axis. Elevated prevalence of gastrointestinal (GI) dysfunction in individuals with ASD suggested that targeting gut may benefit patients with ASD. Lactobacillus plantarum PS128 (PS128) was reported to be a psychobiotic in several animal studies which modulated the levels of neurotransmitters in different brain areas. The current randomized, placebo-controlled trial was conducted to investigate the psychophysiological effects of PS128 in preschool children with ASD.

DETAILED DESCRIPTION:
Emerging evidences support the gut-brain axis and further microbiota-gut-brain axis. Elevated prevalence of gastrointestinal (GI) dysfunction in individuals with ASD suggested that targeting gut may benefit patients with ASD. Lactobacillus plantarum PS128 (PS128) was reported to be a psychobiotic in several animal studies which modulated the levels of neurotransmitters in different brain areas. The current randomized, placebo-controlled trial was conducted to investigate the psychophysiological effects of PS128 in preschool children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill Diagnostic and Statistical Manual of Mental Disorders fifth version (DSM-V) criteria of Autism Spectrum Disorder
* Do not take any other probiotics for at least 3 weeks before and during the study period

Exclusion Criteria:

* Autistic children with other neurodevelopmental disorders or psychiatric diseases
* With a clinically significant chronic medical condition, including; anemia, brain malformations, metabolic diseases, epilepsy, organic gastrointestinal disorders (i.e. gastroesophageal reflux, food allergies, irritable bowel syndrome (IBS)) and Celiac disease
* On anti-fungal, antibiotics, special diet (i.e. gluten-free diet, casein-free diet, high-protein diet, ketogenic diet) and current use of psychiatric medications within the preceding 3 weeks were excluded
* Known allergy to probiotics

Ages: 30 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of anxiety subscale in Children's Behavior Checklist (CBCL)/Achenbach System of Empirically Based Assessment (ASEBA) at week 8 and week 16 | Baseline, week 8 and week 16
  ASEBA for behavioral assessment
Changes from hyperactivity subscale of Attention-Deficit/Hyperactivity Disorder Test (ADHDT) at week 8 and week 16 | Baseline, week 8 and week 16
  Inattention, hyperactive symptoms evaluation

SECONDARY OUTCOMES:
Gastrointestinal symptoms recorded by using GI Severity Index (6-GSI) at week 8 and week 16 | Baseline, week 8 and week 16
  constipation, diarrhea, stool consistency, stool smell, flatulence, and abdominal pain
Change of total scores at week 8 and week 16 from baseline of Changes of Childhood Asperger Syndrome Test (CAST) | Baseline, week 8 and week 16
  CAST for behavioral assessment
Change of total scores at week 8 and week 16 from baseline of Penn Interactive Peer Play Scale, (PIPPS) | Baseline, week 8 and week 16
  PIPPS for communicative and interactive assessment
Change of total scores at week 8 and week 16 from baseline of Social Interaction Assessment Scale | Baseline, week 8 and week 16
  Communicative and interactive assessment
Comparison of Microbiota composition between week 8 and baseline | Baseline and week 8
  Gut and oral microbiota analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Chen MD, Principal Investigator — Department of Pediatric Neurology, MacKay Children's Hospital
Locations (1):
- Department of Pediatric Neurology, MacKay Children's Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No